CLINICAL TRIAL: NCT07136818
Title: From Blueprint to Practice: an Innovative Dynamic 9-Box Grid for Enhancing Exercise Adherence and Aerobic Capacity in Graduate Students
Brief Title: From Blueprint to Practice: An Innovative Dynamic 9-Box Grid Improves Exercise Participation and Aerobic Capacity in Graduate Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hainan Normal University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: AQNU2024110; 21BTY074 (Other Grant/Funding Number: National Social Science Founda)
Record Dates: First submitted 2025-08-08; First posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Improving Low Exercise Engagement; Addressing Sedentary Behaviors; Enhancing Aerobic Capacity; Bridging the Gap Between Exercise Intention and Action

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Weekly Feedback Group (Experimental): Dynamic placement in a 9-grid matrix (based on aerobic capacity + total exercise volume) updated weekly.
  Interventions: Behavioral: Dynamic 9-Square Grid Health Management with Weekly Feedback
- Monthly Feedback Group (Placebo Comparator): Comparison group testing low-frequency feedback.
  Interventions: Behavioral: Dynamic 9-Square Grid Health Management with Monthly Feedback

INTERVENTIONS:
Behavioral: Dynamic 9-Square Grid Health Management with Weekly Feedback — A dual-axis management system categorizing participants into a 3x3 grid based on aerobic capacity (12-min run test) and total exercise volume (smart-device tracked). Includes weekly personalized feedback, tiered exercise prescriptions, and goal recalibration. Arm 1 receives updates every 7 days.
  Arms: Weekly Feedback Group
Behavioral: Dynamic 9-Square Grid Health Management with Monthly Feedback — Identical grid framework as Arm 1 (aerobic capacity + exercise volume assessment), but with monthly (30-day) feedback cycles. Participants receive delayed optimization strategies and tier adjustments once per calendar month, simulating conventional health programs."
  Arms: Monthly Feedback Group

SUMMARY:
This study aims to develop and validate an innovative dynamic 9-square grid management model to improve aerobic capacity (AC) and physical activity participation among graduate students. The model integrates real-time exercise volume (quantified via smart wearable devices) and aerobic capacity (assessed by 12-minute run tests) into a two-dimensional grid, stratifying participants into five tiers for differentiated interventions.

Using a 2 × 3 mixed-design (feedback frequency: weekly vs. monthly; time points: baseline/mid/post-intervention), 32 healthy graduate students are randomized into two groups:

Weekly feedback (dynamic position updates + tailored optimization strategies).

Monthly feedback (position updates at monthly intervals).

Key components include:

Multimodal assessment: Objective exercise metrics (Huawei Band 6), AC (12-min run), psychological scales (Exercise Identity Scale, Self-Efficacy for Exercise Scale).

Tiered intervention: Customized strategies based on grid positioning (e.g., "Star Talent" optimization vs. "Urgent Attention" support).

Primary outcomes: Changes in AC, total exercise volume (TEV), exercise identity, and self-efficacy.

The study seeks to determine whether weekly dynamic feedback outperforms monthly feedback in sustaining behavioral change and enhancing physiological adaptation. Ethical approval was obtained from Anqing Normal University (AQNU2024110).

ELIGIBILITY:
Inclusion Criteria:

* Graduate students aged between 18 and 30 years.
* Completion of the Physical Activity Readiness Questionnaire (PAR-Q) to confirm readiness for exercise.
* Completion of a sociodemographic questionnaire (including age, gender, and education level).
* Confirmation of absence of exercise contraindications (e.g., conditions that may prevent safe participation in physical activity).
* Confirmation of absence of cardiovascular disease.
* Confirmation of absence of recent lower-limb injuries (occurring within the past 3 months or less).
* Confirmation of absence of chest pain symptoms.
* Ability to provide written informed consent for voluntary participation.

Exclusion Criteria:

* Presence of exercise contraindications identified through the PAR-Q or clinical evaluation.
* History or diagnosis of cardiovascular disease (e.g., heart conditions, stroke, or related disorders).
* Recent lower-limb injuries (e.g., fractures, sprains, or surgeries) within the past 3 months.
* Experience of chest pain symptoms (e.g., angina or discomfort during physical exertion).
* Inability to complete the required questionnaires or assessments due to cognitive or language barriers.
* Presence of any uncontrolled chronic condition that could interfere with exercise participation, as determined by the researchers during screening.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2024-10-14 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2025-01-10 (Actual)

PRIMARY OUTCOMES:
Change in Aerobic Capacity (12-min run distance) | Baseline, Week 5 (mid-intervention), Week 9 (post-intervention).
  Description: Distance run in meters during standardized 12-minute field test.
  Measurement Tool: GPS-tracked outdoor run (Keep App + Huawei Band 6).

SECONDARY OUTCOMES:
Exercise Self-Efficacy (SEE-C Scale) | Timeframe: Baseline and Week 9.
  Description: Confidence in maintaining exercise habits (0-90 scale).
  Measurement Tool: Chinese Self-Efficacy for Exercise Scale (Cronbach's α=0.75).

CONTACTS AND LOCATIONS:
Locations (1):
- Hainan Normal University, Haikou, Hainan, China

IPD SHARING:
Plan to Share IPD: Yes
Aerobic capacity test results；Smart wearable exercise data；Cloud-synced TEV metrics (intensity/duration/frequency)；Aggregated weekly values；Psychological scales (EIS/SEE-C)；Encrypted survey responses；Baseline demographics；Limited metadata (age/BMI)。
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 1 January 2030;
Access Criteria: Academic researchers affiliated with accredited institutions Regulatory bodies (e.g., ethics committees) Peer reviewers for journal publication validation
  Access Process:
  Step 1: Submit research proposal via OpenClinica Platform Step 2: Institutional ethics approval documentation required Step 3: Data Use Agreement (DUA) signing with corresponding authors
URL: https://www.openclinica.com

DOCUMENTS (1):
  • Informed Consent Form (2024-09-09): https://cdn.clinicaltrials.gov/large-docs/18/NCT07136818/ICF_000.pdf